CLINICAL TRIAL: NCT05507645
Title: Recombinant Human Prourokinase（rhPro-UK）for Injection Versus Standard Medical Treatment for Acute Mild Ischemic Stroke (NIHSS≤5) Within 4.5 Hours After Symptom Onset
Brief Title: ProUrokinase for Mild Ischemic Cerebrovascular Events (PUMICE)
Acronym: PUMICE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yongjun Wang, professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HX-A-2022032
Record Dates: First submitted 2022-08-17; First posted 2022-08-19 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-07

CONDITIONS: Ischemic Stroke; Mild; Thrombosis
MeSH Terms: conditions — Ischemic Stroke; Lymphoma, Follicular; Thrombosis | interventions — Injections; Aspirin; Clopidogrel; Anticoagulants

STUDY DESIGN:
Intervention Model Description: A multicenter, prospective, randomized, open-label, blinded-endpoint (PROBE) controlled trial
Who Masked: Outcomes Assessor
Masking Description: blinded-endpoint
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- rhPro-UK (35mg) (Experimental): rhPro-UK: 35 mg (5 mg per vial, 7 vials in total) Dissolve 15mg (3 vials) of rhPro-UK in 10ml of saline and intravenous bolus within 3 minutes, and dissolve the remaining 20mg (4 vials) in 90ml of saline and intravenous drip within 30 minutes. (Note: after adding saline, overturn it gently once to twice, do not shake vigorously, so as to avoid foaming of the rhPro-UK solution and reduce the efficacy).
  Interventions: Drug: Recombinant Human Prourokinase for Injection (rhPro-UK)
- standard medical treatment (Active Comparator): Standard antiplatelet or anticoagulant treatment at the discretion of local investigators according to the 'Chinese guidelines for diagnosis and treatment of acute ischemic stroke 2018'.
  Interventions: Drug: standard medical treatment

INTERVENTIONS:
Drug: Recombinant Human Prourokinase for Injection (rhPro-UK) — 15mg of rhPro-UK intravenous bolus within 3 minutes, and the remaining 20mg intravenous drip within 30 minutes.
  Other Names: Puyouke
  Arms: rhPro-UK (35mg)
Drug: standard medical treatment — Standard antiplatelet or anticoagulant treatment at the discretion of local investigators.
  Other Names: Aspirin, clopidogrel, anticoagulant
  Arms: standard medical treatment

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of rhPro-UK (35mg) versus standard medical treatment in acute mild ischemic stroke within 4.5 hours of symptom onset.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, patients who meet the eligibility requirements will be randomized to recombinant human Prourokinase for injection (rhPro-UK) or standard medical treatment in a 1:1 ratio. Written informed consent will be needed.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, any gender;
2. Acute ischemic stroke symptom onset within 4.5 hours prior to enrollment; onset time refers to 'last-seen normal time';
3. Pre-stroke mRS score≤ 1;
4. Baseline NIHSS ≤ 5 (both included);
5. Written informed consent from patients or their legally authorized representatives

Exclusion Criteria:

1. Rapidly improving symptoms at the discretion of the investigator;
2. Intended to proceed to endovascular treatment during 90 days (including mechanical thrombectomy, stent insertion or balloon expansion);
3. Allergy to rhPro-UK and it's components (human albumin, mannitol);
4. NIHSS consciousness score 1a >2, or epileptic seizure, hemiplegia after seizures (Todd's palsy) or combined with other nervous/mental illness unable to cooperate or unwilling to cooperate;
5. Persistent blood pressure elevation (systolic ≥180 mmHg or diastolic ≥100 mmHg), despite blood pressure lowering treatment;
6. Blood glucose <2.8 or >22.2 mmol/L (point of care glucose testing is acceptable);
7. Active internal bleeding or at high risk of bleeding, e.g.: Major surgery, trauma or gastrointestinal or urinary tract haemorrhage within the previous 21 days, or arterial puncture at a non-compressible site within the previous 7 days;
8. Any known impairment in coagulation due to comorbid disease or anticoagulant use. If on warfarin, then INR >1.7 or prothrombin time >15 seconds; if use of any direct thrombin inhibitors or direct factor Xa inhibitors or new oral anticoagulants (NOAC) during the last 48 hours unless reversal of effect can be achieved with a reversal agent (by idarucizumab) or sensitivity laboratory test values greater than the upper limit of normal (eg, activated partial thromboplastin time (aPTT), international normalized ratio (INR), platelet count, thrombin time (TT), or appropriate factor Xa activity assay); if on any full dose heparin/heparinoid during the last 24 hours or with an elevated aPTT greater than the upper limit of normal;
9. Known defect of platelet function or platelet count below 100,000/mm3 (but patients on antiplatelet agents can be included);
10. Ischemic stroke or myocardial infarction in previous 3 months, previous intracranial haemorrhage, severe traumatic brain injury or intracranial or intraspinal operation in previous 3 months, or known intracranial neoplasm (except for neuroectodermal tumors, such as meningiomas), arteriovenous malformation or giant aneurysm;
11. Any terminal illness such that patient would not be expected to survive more than 1 year
12. Large cerebral infarction (infarct size > 1/3 MCA territory) on CT or MRI;
13. Acute or past intracerebral hemorrhage (ICH) identified by CT or MRI (including intraparenchymal hemorrhage, intraventricular hemorrhage, subarachnoid hemorrhage, subdural/epidural hematoma);
14. Pregnant women, nursing mothers, or reluctant to agree taking effective contraceptive measures during the period of trial subjects;
15. Any condition that, in the judgment of the investigator could impose hazards to the patient if study therapy is initiated or affect the participation of the patient in the study;
16. Participation in other interventional clinical trials within the previous 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1446 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2024-03-26 (Actual); Study Completion 2024-06-17 (Actual)

PRIMARY OUTCOMES:
The modified Rankin Scale score (mRS) ≤ 1 at 90 days | 90 days
  The proportion of the modified Rankin Scale score (mRS) ≤ 1 at 90 days.

SECONDARY OUTCOMES:
Ordinal distribution of mRS at 90 days | 90 days
  Ordinal distribution of mRS at 90 days
mRS score ≤ 2 at 90 days | 90 days
  The proportion of mRS score ≤ 2 at 90 days
Early neurological functional improvement | 24 hours
  Clinical response rate at 24 hours defined as an improvement on NIHSS score ≥ 4 points compared with the initial deficit or NIHSS score ≤ 1 point
Barthel index of 75-100 points at 90 days | 90 days
  The proportion of Barthel index of 75-100 points at 90 days
Quality of Life (EQ-5D-5L) at 90 days | 90 days
  The value of Quality of Life (EQ-5D-5L) at 90 days
Activities of Daily Living (Lawton IADL) at 90 days | 90 days
  The score of Activities of Daily Living (Lawton IADL) at 90 days
Symptomatic intracranial hemorrhage within 36 hours | 36 hours
  The rate of symptomatic intracranial hemorrhage within 36 hours (as defined by ECASS III)
All-cause death at 90 days | 90 days
  All-cause mortality at 90 days
Systematic bleeding at 90 days | 90 days
  The rate of systematic bleeding at 90 days (as defined by GUSTO: moderate and severe bleeding)
Adverse events (AEs)/ serious adverse events (SAEs) within 90 days | 90 days
  The proportion of AEs/SAEs within 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Yongjun Wang, MD, Principal Investigator — Beijing Tiantan Hospital
Locations (89):
- China (89):
  - Taihe Hospital of Traditional Chinese Medicine, Fuyang, Anhui
  - Lujiang County People's Hospital,Anhui Province, Hefei, Anhui
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The First Hospital of Fangshan District, Beijing, Beijing, Beijing Municipality
  - Chongqing Sanbo Chang 'an Hospital, Chongqing, Chongqing Municipality
  - Dingxi People's Hospital, Dingxi, Gansu
  - Jiuquan City People's Hospital, Jiuquan, Gansu
  - Guangdong Second Provincial General Hospital, Guangzhou, Guangdong
  - Heyuan People's Hospital, Heyuan, Guangdong
  - People's Hospital of Huazhou, Maoming, Guangdong
  - Wuchuan People's Hospital, Zhanjiang, Guangdong
  - Wuming Hospital of Guangxi Medical University, Nanning, Guangxi
  - The Second People's Hospital of Guiyang, Guiyang, Guizhou
  - The Second Affiliated Hospital of Guizhou Medical University, Kaili, Guizhou
  - The People's Hospital of the Qiandongnan Miao and Dong Autonomous Prefecture, Kaili, Guizhou
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - Hebei Tang County People Hospital, Baoding, Hebei
  - Chengde Central Hospital, Chengde, Hebei
  - Long Hua Xian Yi Yuan, Chengde, Hebei
  - Fengning Manchu Autonomous County Hospital, Chengde, Hebei
  - Wei Xian Ren Min Yi Yuan, Handan, Hebei
  - The People's Hospital of Changli County, Qinhuangdao, Hebei
  - The Second Hospital of Qinhuangdao, Qinhuangdao, Hebei
  - Xingtang People's Hospital, Shijiazhuang, Hebei
  - Yuanshi Hospital of Traditional Chinese Medicine, Shijiazhuang, Hebei
  - The Second Hospital of Xinji, Shijiazhuang, Hebei
  - Xinji Hospital of T.C.M, Shijiazhuang, Hebei
  - Linxi Hospital of Kailuan General Hospital, Tangshan, Hebei
  - Luanzhou People's Hospital, Tangshan, Hebei
  - Tangshan Guye Traditional Chinese Medicine Hospital, Tangshan, Hebei
  - Tangshan Fengnan District Hospital, Tangshan, Hebei
  - Yu Tian Xian Zhong Yi Yi Yuan, Tangshan, Hebei
  - Zunhua People's Hospital, Tangshan, Hebei
  - The People's Hospital of Qianxi County, Tangshan, Hebei
  - Weixian People's Hospital, Xingtai, Hebei
  - The Greatwall Hospital, Xingtai, Hebei
  - Center Hospital·Jiamusi, Jiamusi, Heilongjiang
  - Central Hospital·Jiaozuo, Jiaozuo, Henan
  - The Second People's Hospital of Jiaozuo, Jiaozuo, Henan
  - Jiyuan Hospital of Traditional Chinese Medicine, Jiyuan, Henan
  - Luoyang First People's Hospital, Luoyang, Henan
  - Tanghe County People's Hospital, Nanyang, Henan
  - Puyang Oilfield General Hospital, Puyang, Henan
  - Chinese Medicine Hospital of Puyang, Puyang, Henan
  - The First People Hospital of Lingbao, Sanmenxia, Henan
  - The Shangqiu First People's Hospital, Shangqiu, Henan
  - Xiayi County People's Hospital, Shangqiu, Henan
  - The People's Hospital of Yongcheng, Shangqiu, Henan
  - People's Hospital of Xixian, Xinyang, Henan
  - Guang Shan County People's Hospital, Xinyang, Henan
  - Xinmi Hospital of T.C.M, Zhengzhou, Henan
  - Taikang Xian People's Hospital, Zhoukou, Henan
  - Liuyang Jili Hospital, Changsha, Hunan
  - Baotou City Central Hospital, Baotou, Inner Mongolia
  - Huai'an Second People's Hospital, Huai'an, Jiangsu
  - Funing People's Hospital, Yancheng, Jiangsu
  - Jilin People's Hospital, Jilin, Jilin
  - Tonghua City vascular disease Hospital and Dongchang District People's Hospital, Tonghua, Jilin
  - Meihekou Central Hospital, Tonghua, Jilin
  - Haicheng Hospital of T.C.M, Anshan, Liaoning
  - Dalian Lvshunkou District Traditional Chinese Medicine Hospital, Dalian, Liaoning
  - General Hospital of Fushun Mining Bureau of Liaoning Health Industry Group, Fushun, Liaoning
  - Huludao Center Hospital, Huludao, Liaoning
  - The Second People's Hospital of Huludao, Huludao, Liaoning
  - The Fourth Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Weinan Central Hospital, Weinan, Shaanxi
  - People's Hospital of Qihe County, Dezhou, Shandong
  - Ningjin People's Hospital, Dezhou, Shandong
  - Liaocheng People's Hospital, Liaocheng, Shandong
  - Liaocheng Third People's Hospital, Liaocheng, Shandong
  - Guanxian People's Hospital, Liaocheng, Shandong
  - The People's Hospital of Gaotang, Liaocheng, Shandong
  - People's Hospital of Yinan, Linyi, Shandong
  - The Second Affiliated Hospital of Shandong First Medical University, Tai’an, Shandong
  - Weihai Central Hospital, Weihai, Shandong
  - Weihai Wendeng District People's Hospital, Weihai, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Yantai Taocun Central Hospital, Yantai, Shandong
  - Qixia Traditional Chinese Medicine Hospital, Yantai, Shandong
  - Zibo Central Hospital, Zibo, Shandong
  - Zibo Municipal Hospital, Zibo, Shandong
  - Shanghai Putuo Liqun Hospital, Shanghai, Shanghai Municipality
  - Linfen Central Hospital, Linfen, Shanxi
  - Yangquan Coal Industry(Group) General Hospital, Yangquan, Shanxi
  - Yangquan First People's Hospital, Yangquan, Shanxi
  - Affiliated Hospital of North Sichuan Medical College, Nanchong, Sichuan
  - People's Hospital of Yilong County, Nanchong, Sichuan
  - Suining Central Hospital, Suining, Sichuan
  - Tianjin 4th Center Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xiong Y, Meng X, Jin A, Campbell BCV, Xu A, Dong Q, Xu Y, Pan Y, Jiang Y, Niu S, Li Z, Zhuang X, Guo N, Yuan Z, Kong Z, Zong L, Duan C, Cao Z, Wang L, Hao M, Wu S, Feng X, Li H, Wu N, Li Z, Zhao X, Wang Y; PUMICE Investigators. Prourokinase vs Standard Care for Patients With Mild Ischemic Stroke: The PUMICE Randomized Clinical Trial. JAMA Neurol. 2025 Mar 1;82(3):258-266. doi: 10.1001/jamaneurol.2024.4688. PMID 39836393
- [Derived] Xiong Y, Hao M, Pan Y, Duan C, Feng X, Li H, Wu N, Wang L, Meng X, Zhao X, Wang Y; PUMICE investigators*. Rationale and design of ProUrokinase in Mild IsChemic strokE (PUMICE): a multicentre, prospective, randomised, open-label, blinded-endpoint controlled trial. Stroke Vasc Neurol. 2024 Dec 30;9(6):715-722. doi: 10.1136/svn-2023-002673. PMID 38296588